CLINICAL TRIAL: NCT02271867
Title: Thermal Quantitative Sensory Testing as a Method to Semi-quantitatively Assess the Neurosensory Effects of 3 Local Anesthetic Solutions in an Interscalene Block
Brief Title: Thermal QST for Interscale Block Evaluation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Ethisch Comité UZ Antwerpen, Thermal Quantitative Sensory Testing as a method to semi-quantitatively assess the neurosensory effects of 3 local anesthetic solutions in an interscalene block, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: EC 9/25/113
Record Dates: First submitted 2014-10-13; First posted 2014-10-22 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Anesthetics, Local; Nerve Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Levobupivacaine 0,5% (Active Comparator): Levobupivacaine 0,5% 15 ml once
  Interventions: Procedure: Interscalene block
- Levobupivacaine 0,5% with epinephrine (Active Comparator): Levobupivacaine 0,5% with 1/200000 epinephrine 15 ml once
  Interventions: Procedure: Interscalene block
- Ropivacaine 0,75% (Active Comparator): Ropivacaine 0,75% 15 ml once
  Interventions: Procedure: Interscalene block

INTERVENTIONS:
Procedure: Interscalene block — An ultrasound guided ISB was performed with injection aimed to block the C5-root

SUMMARY:
Thermal quantitative sensory testing (QST) is a method to evaluate peripheral nerve blocks in a quantitative way. It assesses the neurosensory effects of local anesthetics, like nerve block intensity, duration, recovery, neurotoxicity, the effect of spread of local anesthetic solutions and the effect and the eventual neurotoxicity of adjuvants. We aimed at investigating, in a quantitative way, the block characteristics of 3 different commonly used local anesthetics on peripheral nerves through the application of thermal QST by measuring changes in sensory detection thresholds. Furthermore, we wanted to evaluate if QST could be of value for measuring gradual changes in block characteristics on the adjacent nerves at distance of the injection site in an US-ISB.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for diagnostic and therapeutic shoulder arthroscopy, with or without decompression technique were eligible

Exclusion Criteria:

* contraindications for ISB
* diabetes mellitus
* peripheral neuropathy
* patients receiving chronic analgesic therapy
* contraindications for NSAID
* patients with an initial QST with abnormal values

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-07; Primary Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Presence of sensory block | 24 hours after intervention

SECONDARY OUTCOMES:
Degree of sensory stimulus detection threshold variation from baseline values | 24 hours after intervention
  The higher the difference in detection threshold variation, the more intense the block. Measured as % change, where 100% change means no sensation on maximal QST stimulus (0°C for cold sensation and 50°C for warm sensation)
Block duration | 24 hours after intervention
Use of rescue medication | 24 hours after intervention
Presence of motor block | 24 hours after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

REFERENCES:
- [Derived] Sermeus LA, Hans GH, Schepens T, Bosserez NM, Breebaart MB, Smitz CJ, Vercauteren MP. Thermal quantitative sensory testing to assess the sensory effects of three local anesthetic solutions in a randomized trial of interscalene blockade for shoulder surgery. Can J Anaesth. 2016 Jan;63(1):46-55. doi: 10.1007/s12630-015-0505-x. Epub 2015 Oct 16. PMID 26475166